CLINICAL TRIAL: NCT05447520
Title: Clinical Study Evaluating the Efficacy and Safety of Adjunctive Use of Montelukast in Rheumatoid Arthritis Patients
Brief Title: Montelukast Use in Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Noha Mansour (Other)
Responsible Party: Sponsor-Investigator, Noha Mansour, Principal investigator-Lecturer of Clinical Pharmacy-Clinical Pharmacy and Pharmacy Practice Department, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2021-376
Record Dates: First submitted 2022-07-01; First posted 2022-07-07 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Montelukast Group (Experimental): Patients will receive conventional DMARDs plus montelukast 10 mg tablet once daily for 16 weeks.
  Interventions: Drug: Montelukast; Drug: Conventional DMARDs
- Control Group (Placebo Comparator): Patients will receive conventional DMARDs plus placebo tablet daily for 16 weeks
  Interventions: Drug: Placebo; Drug: Conventional DMARDs

INTERVENTIONS:
Drug: Montelukast — Montelukast 10 mg oral tablet once daily for RA patients with moderate to high disease activity provided by DAS-28 score greater than 3.2
  Arms: Montelukast Group
Drug: Placebo — Oral tablet once daily
  Arms: Control Group
Drug: Conventional DMARDs — methotrexate, leflunomide, hydroxychloroquine or sulfasalazine

SUMMARY:
Montelukast is widely used in patients with asthma. Several preclinical data suggest that it could be repositioned as novel strategy for managing rheumatic patients by decreasing inflammatory mediators.

Considering the probable enhanced antiarthritic effects of montelukast; it could be hypothesized that its adjuvant use might improve treatment outcomes in rheumatic patients who remain poorly controlled despite initial optimal guidelines directed medical treatment. Therefore, this study aims to evaluate the potential added benefits of montelukast use in conjunction with csDMARDs in RA patients with moderate and high disease activity.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ages ≥ 18 years old.
* Patients diagnosed with RA according to American College of Rheumatology/European league Against Rheumatism (ACR/ EULAR) 2010 criteria (25) presented with disease activity score-28 based on C-reactive protein (CRP) levels (DAS-28-CRP) >3.2.
* Patient received stable regimen of one or more csDMARDs for at least the past 3 months.

Exclusion Criteria:

* Patient taking biological DMARDs.
* Known hypersensitivity to montelukast.
* Patients receive montelukast for any other indications.
* Patients with impaired liver functions (liver transaminases level ≥ three times upper normal limits).
* Patients with impaired kidney (estimated glomerular filtration rate (eGFR) < 30 ml/min).
* Pregnancy and lactation.
* Patients with active or severe infections.
* Patients with other inflammatory or autoimmune diseases and malignancies.
* Patients with any psychiatric disorder.
* Patients taking IV, IM, orally (dose > 10 mg daily) or intra articular corticosteroides,
* Smokers.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Disease activity score in 28 joints (DAS-28) | 16 weeks
  Scale assessing severity of rheumatoid arthritis based on number of tender , swollen joints , CRP levels ,and patient self-assessment of his condition (global health assessment) . Whereas "28" describes the number of different joints including in the measurement :proximal interphalangeal joints (10 joints),metacarpophalangeal joints (10),wrists (2),elbows (2),shoulders (2),knees (2).
  A DAS-28 value < 2.6 corresponds to remission,value between 2.6 and 3.2 corresponds to a low disease activity, value between 3.2 and 5.1 corresponds to a moderate disease activity, and DAS28 value >5.1 corresponds to a high disease activity.

SECONDARY OUTCOMES:
Assessment of patient's QOL using Health Assessment Questionnaire Disability index (HAQ-DI) | 16 weeks
  It comprises eight categories assessing the ability of patients to perform activities of daily living. Each category includes two or three questions scored from 0 (without any difficulty) to 3 (unable to do).
  * The score of each category is the highest score among the scores of the included questions.
  * If an aid or assistance device is used or if help is required from another individual, then the minimum score for that section is 2.
  * The final score is calculated by summation of the scores for various categories divided by the number of categories.
  * Resulting in a score from 0 to 3.

CONTACTS AND LOCATIONS:
Overall Officials: Noha Mansour, Principal Investigator — Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Egypt